CLINICAL TRIAL: NCT00671502
Title: Randomized, Double-Blind, Double-Dummy Trial of Two Sustained Release Formulations of Carisoprodol Compared to Placebo in Subjects With Acute, Painful, Musculoskeletal Spasm of the Lower Back
Brief Title: A Study to Evaluate Two Formulations of Carisoprodol in Subjects With Musculoskeletal Spasm of the Lower Back
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP510
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Results first posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-10

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Carisoprodol; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carisoprodol 700mg (Experimental): tablet sustained release (SR)
  Interventions: Drug: Carisoprodol SR
- Carisoprodol 500mg (Experimental): sustained release(SR) tablet
  Interventions: Drug: Carisoprodol SR
- Placebo (Placebo Comparator): tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carisoprodol SR — 700 mg twice daily
  Other Names: sustained release(SR)
  Arms: Carisoprodol 700mg
Drug: Carisoprodol SR — 500 mg twice daily
  Other Names: sustained release(SR) tablet
  Arms: Carisoprodol 500mg
Drug: Placebo — Placebo tablet
  Other Names: no other name
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if two sustained released formulations of carisoprodol are more effective than placebo.

DETAILED DESCRIPTION:
Methodology:

This was a randomized, double-blind, double-dummy, placebo-controlled, parallel-group study in subjects 18-70 years of age with acute, painful, muscle spasm of the lower back. The study consisted of a baseline screening (Study Day 1), during which subjects were evaluated for inclusion/exclusion criteria, and a 7-day double-blind treatment period (Study Day 1 through Study Day 7). Subjects were randomly assigned to be dosed twice daily with one of the following double-blind treatments: sustained release(SR) carisoprodol 500-mg tablets,sustained release (SR) carisoprodol 700-mg tablets, or placebo.

Subjects were evaluated in the clinic on Study Days 1, 3 and 7. Subjects who remained symptomatic on Study Day 7 were allowed to continue in the study for a 7-day, double-blind extension period at the discretion of the Investigator. Subjects were contacted by telephone for a safety follow-up 7 days after the last dose of study medication.

A pharmacokinetic (PK) substudy was conducted at selected sites. These sites obtained blood samples for PK analysis at the end of the 7-day treatment period and the 14-day treatment period, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Onset of pain is within 3 days of first visit
* Subject rating of pain must be 40 mm or greater on visual analog scale( VAS)
* Ability to discontinue all analgesics, non steroidal anti inflammatory drug (NSAIDs), and other muscle relaxants
* Willingness to provide written informed consent
* Must be in generally good health

Exclusion Criteria:

* Presence of sciatic pain
* History of clinically significant spine pathology such as herniated nucleas pulposis, spondylolisthesis, spinal stenosis
* Presence of underlying chronic back pain
* Neurological signs and symptoms such as numbness, tingling, foot drop, parethesia, unexplained constipation, urinary retention or urinary incontinence
* Myocardial infaction within one year of study
* Cancer not in remission or in remission less than one year
* HIV or other immunodeficiency syndromes
* History of osteoporosis or at high risk for vetebral fracture
* Underlying rheumatologic disease such as rheumatoid arthritis, ankylosing spondylitis, etc.
* Presence of active influenze or other viral syndromes
* Morbid obesity basal metabolic index(BMI >39)
* Evidence of infection, such as low grade fever or neutrophilia
* Existence of any medical/surgical condition that could interfere with the evaluation of the study medication
* Known history of alcohol or drug abuse
* Injury involving high potential for litigation, including worker's compensation or automobile accidents
* Pregnancy or breast feeding
* Women of child-bearing potential not abstinent or not practicing a medically acceptable method of contraception
* Vertebral body or spinous process, percussive tenderness on physical exam
* Any abnormalities in the following tests of both lower extremities: ankle dorsiflexion strength, great toe dorsiflexion strength, absent or hypereflexic Achilles or patellar tendor reflexes, abnormal sensory exam in the medial, dorsal or lateral aspect of the foot and positive straight leg raise test
* Urgent medical conditions on comprehensive exam that might indicate a more serious condition should be treated urgently

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M. Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (68):
- United States (68):
  - MedSearch, LLC, Birmingham, Alabama
  - Genesis Clinical Research Corporation, Huntsville, Alabama
  - Vaughn H. Mancha, Jr., PC Family Practice, Montgomery, Alabama
  - Anasazi Internal Medicine PC, Phoenix, Arizona
  - Heritage Physician Group, Hot Springs, Arkansas
  - OrthoArkansas, Little Rock, Arkansas
  - Family Practice Clinic, North Little Rock, Arkansas
  - Quality of Life Medical Center, LLC, Hawaiian Gardens, California
  - Trinity Health and Wellness, Roseville, California
  - San Diego Sports Medicine & Family Health Center, San Diego, California
  - Quality Care Medical Center, Inc., Vista, California
  - Anthony Roselli, MD, Avon, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - Southeastern Integrated Medical, PL dba Florida Medical Research Institute, Gainesville, Florida
  - South Florida Clinical Research Center, Hollywood, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Genesis Research International, Longwood, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Tukoi Clinical Research, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Sunrise Medical Research #501, Plantation, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Perimeter Institute for Clinical Research, Inc., Atlanta, Georgia
  - Sunset Medical Research, Sunset, Louisiana
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Northern Pines Health Center, Buckley, Michigan
  - KMED Research, Clair Shores, Michigan
  - Harris & Associates, P.C., Detroit, Michigan
  - Valley Medical Center, Flint, Michigan
  - Westside Family Medical Center, P.C., Kalamazoo, Michigan
  - Kansas City University of Medicine and BioSciences Dybedal Building, Kansas City, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - South Jersey Medical Associations, PA, Blackwood, New Jersey
  - Care Center of Family Practice & Pediatrics of Hamilton, Hamilton, New Jersey
  - Partners in Primary Care, Voorhees Township, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Metrolina Medical Research, Charlotte, North Carolina
  - Clinical Research Source Inc., Perrysburg, Ohio
  - Family Practice Center of Wadsworth, Inc., Wadsworth, Ohio
  - Integrated Medical Research, Ashland, Oregon
  - Williamette Valley Clinical Studies, Eugene, Oregon
  - Fanno Creek Clinic, LLC, Portland, Oregon
  - Best Clinical Research - PA, Philadelphia, Pennsylvania
  - Arcuri Clinical Research, Philadelphia, Pennsylvania
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Robert S. Eagerton Jr., MD Family Practice, Manning, South Carolina
  - Holston Medical Group, P.C., Bristol, Tennessee
  - ACRC Trials, Addison, Texas
  - Arlington Family Health Pavilion, Arlington, Texas
  - Central TX Clinical Research, Austin, Texas
  - Mid-Cities Family Care, Bedford, Texas
  - Evergreen Clinical Research, LLC, Bellaire, Texas
  - Deer Park Family Clinic, P.A., Deer Park, Texas
  - Prime Care Medical Group, Houston, Texas
  - West Houston Clinical Research, Houston, Texas
  - North Hills Family Practice, North Richland Hills, Texas
  - North Texas Family Medicine, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Unlimited Research, San Antonio, Texas
  - InVisions Consultants, LLC, San Antonio, Texas
  - Oakwell Clinical Research, San Antonio, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Medical Research Initiatives, Richmond, Virginia
  - Liberty Research Center, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Carisoprodol 700mg; Carisoprodol 500mg Tablet: tablet experimental formulation
- Placebo Tablet: tablet placebo no experimental formulation
Period: Overall Study
Arm/Group | Carisoprodol 700mg | Carisoprodol 500mg Tablet | Placebo Tablet
Started | 281 | 280 | 279
Completed | 242 | 241 | 252
Not Completed | 39 | 39 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carisoprodol 700mg | Carisoprodol 500mg Tablet | Placebo Tablet | Total
Number analyzed (Participants) | 281 | 280 | 279 | 840
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 278 | 278 | 275 | 831
  >=65 years | 3 | 2 | 4 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 40.3 (13.05) | 41.4 (12.6) | 40.9 (12.72) | 40.9 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 144 | 136 | 413
  Male | 148 | 136 | 143 | 427
Region of Enrollment [Number; unit: participants]
  United States | 281 | 280 | 279 | 840

OUTCOME MEASURES:

1. Primary Outcome: Subject Rating of Pain on a 100-point Visual Analog Scale (VAS)
Description: the scale used was from 0 to 100 mm. 0 equaled no pain and 100 equaled maximum pain.participants measure their pain before treatment and during treatment at each visit
Time Frame: up to 14 days
Population: efficacy analyses based on ITT population. LOCF used to impute missing data. To detect a 14% difference between the carisoprodol and placebo treated subjects, 196 ITTsubjects per group (alpha level 0.025,power 80%).Assuming 15% dropout rate, 226 subjects per group were needed.A total of678 subjects were required to achieve 584 ITT subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Groups:
- Carisoprodol 500mg Tablets: carisoprodol 500mg tablets treatment arm
- Carisoprodol 700mg Tablets: carisoprodol 700mg tablets treatment arm
- Placebo Tablets: placebo tablets treatment arm
Arm/Group | Carisoprodol 500mg Tablets | Carisoprodol 700mg Tablets | Placebo Tablets
Number analyzed (Participants) | 280 | 281 | 279
mm | 27.5 [-21 to 83] | 28 [-19 to 89] | 28.6 [-36 to 82]

2. Secondary Outcome: Subject Functional Assessment Based on the Roland-Morris Disability Questionnaire (RMDQ)
Time Frame: up to 14 days
Reporting Status: Not Posted

3. Secondary Outcome: Adverse Event Assessment
Description: the number of adverse events reported during the course of the study as reported by the participants
Time Frame: up to 21 days
Reporting Status: Not Posted
Measure: Number; unit: participants

ADVERSE EVENTS:
Time Frame: up to 21 days
Arm/Group | Carisoprodol 700mg | Carisoprodol 500mg Tablet | Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 0/278 | 1/280 | 0/275
Other Adverse Events (participants affected / at risk) | 78/278 | 65/280 | 37/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carisoprodol 700mg (N=278) | Carisoprodol 500mg Tablet (N=280) | Placebo Tablet (N=275)
transient ischemic attack (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — occurred after discontinuation of drug therefore not considered treatment emergent
OTHER ADVERSE EVENTS (reported when occurring in more than 0.7% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Carisoprodol 700mg (N=278) | Carisoprodol 500mg Tablet (N=280) | Placebo Tablet (N=275)
somnolence (Nervous system disorders) | 44/44 (44) | 36 (36) | 18 (18)
dizziness (Nervous system disorders) | 23 (23) | 12 (12) | 6 (6)
nausea (Gastrointestinal disorders) | 5 (5) | 12 (12) | 6 (6)
fatigue (General disorders) | 5 (5) | 5 (5) | 2 (2)
headache (General disorders) | 8 (8) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No